CLINICAL TRIAL: NCT05810467
Title: Active Surveillance Study for Prostate Cancer Management for Men at Higher Genetic Risk Compared With Men at No Known Higher Genetic Risk.
Brief Title: The Active Surveillance Study
Acronym: AS
Status: Recruiting | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other); North Bristol NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5747
Record Dates: First submitted 2023-03-21; First posted 2023-04-12 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — This study will look at the association of biomarkers with PrCa presentation and progression among men on Active Surveillance and stratify it by their genetic risk. It will also investigate the incidence and progression by differing genetic risks. The study will review serial PSA, biomarkers and imaging data for men in AS comparing and contrasting those of known higher genetic risk for PrCa with those without a known higher genetic risk. Samples will be collected to investigate the association of genetic profiles and biomarkers from biological samples including plasma, serum, urine, stool, and saliva in these two groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Arm: Men diagnosed with low-grade PrCa undergoing Active Surveillance and are not known to have an increased genetic risk for PrCa e.g. Men without high-risk mutations or high polygenic risk score (PRS).
  Men diagnosed with PrCa suitable for Active Surveillance who wish to continue follow up at collaborating hospitals will be offered enrolment in collection and monitoring of various biological samples. These men will act as a control group, as they do not have a known higher genetic risk of PrCa. The control group will have genetic analysis carried out on provided saliva or blood samples. Their family history will be captured. They will be genotyped using the latest technology and at a minimum have PRS testing done.
  Men may be moved out of the control arm and into the high-risk arm, if identified at a higher genetic risk or as having a strong family history of PrCa for the purposes of the analysis. Any clinically significant genetic results will be discussed with the participants.
  Interventions: Other: Active Surveillance
- High-risk Arm: Men who have been diagnosed with low grade PrCa and are undergoing active surveillance who are at genetically higher risk of PrCa defined as:
  1. Men of any ancestry with a family history defined as at least one first degree (or second degree if through the female line) relative with PrCa diagnosed at <70 years (diagnosis verified).
  2. Men of Black African or Caribbean ancestry irrespective of family history
  3. Men of any ancestry known to carry a mutation in a high-risk gene thought to cause a higher risk of prostate cancer.
  4. Men of ancestry with a high genetic risk (common and/or rare variants) for prostate cancer resulting in relative risk (RR) of ≥2.
  Interventions: Other: Active Surveillance

INTERVENTIONS:
Other: Active Surveillance — Active surveillance (AS) is an accepted management strategy for men diagnosed with low risk PrCa, generally defined as PSA <10ng/ml and Gleason score of ≤6 and clinical stage T1 to T2a. Occasionally, a minority of men with Gleason 3+4 disease are included, though majority of those included in AS studies have Gleason 3+3 disease or less.
  Men in AS studies have repeated biopsies based on various criteria including PSA velocity, repeat biopsy at set time points and change noted on digital rectal examination (DRE), biopsy or MRI imaging. Progression of disease has been defined in various ways in different studies, generally, using criteria of Gleason upgrade to greater than Gleason 3+3, evidence of Gleason 4 or Gleason 5 disease, >50% involvement of any one biopsy core, and greater than 2 cores positive on repeat biopsy. Percentages of men on AS who have upgrade on repeat biopsy have been found to be 19-34%; this may differ in our cohort of men with increased genetic risk for PrCa.

SUMMARY:
The Active Surveillance study is a prospective study developed to look at the association of biomarkers with PrCa presentation and progression among men on Active Surveillance and stratify it by their genetic risk. This study will also investigate the incidence and progression by differing genetic risks.

DETAILED DESCRIPTION:
This prospective study will look at the association of biomarkers with PrCa presentation and progression among men on Active Surveillance and stratify it by their genetic risk. This study will also investigate the incidence and progression by differing genetic risks. The study will review the serial PSA and imaging data for men in AS comparing and contrasting the men of known higher genetic risk for PrCa with those without a known higher genetic risk. Additionally, the study aims to collect samples to investigate the profile of plasma, serum, urine, stool, and saliva (or DNA from blood) biomarkers in men at a higher genetic risk of PrCa, who have been diagnosed with low risk PrCa and are undergoing Active Surveillance. It will also review the association of specific genetic profiles and biomarkers (biological samples - plasma, serum, urine, stool and saliva - where possible, DNA from blood will be used instead of saliva samples). These markers will be compared and contrasted with samples from men with no known increased genetic risk for PrCa.

The study aims to recruit a total of 200 men with low grade PrCa, aged ≥18 into two cohorts (i.e. men on AS who are known to be at higher genetic risk and those on AS with no known increased genetic risk of PrCa. Patients will be identified through urology clinics at the Royal Marsden Hospital and North Bristol NHS Trust. These will be men who are already registered at either the Royal Marsden Hospital or North Bristol NHS Trust and undergoing active surveillance (as determined by the MDT) will be given a patient information sheet. This explains the study in lay terms and gives the contact details for the relevant research team.

ELIGIBILITY:
Inclusion Criteria

* Men ≥18 years old under the care of an Active Surveillance clinic.
* Known diagnosis of PrCa, deemed suitable for Active surveillance at multi-disciplinary meeting (MDT).
* Men at genetically higher PrCa risk who are either:

  (1) Men of any ancestry with a positive family history of PrCa defined as:
* Having a first degree relative (or second degree if through female line) with histologically or death certificate proven PrCa diagnosed at <70 years
* Having two relatives on the same side of the family with histologically or death certificate proven PrCa where at least one is diagnosed at <70 years
* Having three relatives on the same side of the family with histologically or death certificate proven PrCa diagnosed at any age

Or (2) Men of Black African or Black African-Caribbean ancestry defined as:

* Both parents and all 4 grandparents from that origin Or (3) Men of any ancestry with a pathogenic mutation in a gene thought to cause a higher risk of prostate cancer: (including BRCA1, BRCA2, ATM, PALB2, MLH1, MSH2, MSH6, CHEK2 and other DNA repair gene mutations as listed in appendix A) Or (4) Men of any ancestry with a high genetic risk (common and/or rare variants) for PrCa resulting in a RR of ≥2 of PrCa
* Men of any ancestry with no known high risk genetic factors who have been diagnosed with low grade PrCa and deemed suitable for Active Surveillance at multi-disciplinary meeting (control group) as defined in the 4 criteria above.
* Who performance status 0-2
* Absence of any psychological, familial, sociological, or geographical situation potentially hampering compliance with the study protocol and follow-up schedule.

Exclusion Criteria

* No PrCa diagnosis
* PrCa diagnosis that is not deemed suitable for active surveillance at multi-disciplinary meeting
* Any significant psychological conditions that may be worsened or exacerbated by participation in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Assigned male at birth.
Study Population: * Control group (i.e., no known high PrCa risk): 100 men
  * Men at genetically higher PrCa risk: 100 men
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To determine the incidence of disease progression of PrCa in the cohorts studied. | The full analysis being completed within one year of date of completion of 5 year follow-up of the last participant.
  Descriptive statistics will be used to determine and compare the characteristics of cancers in each cohort at recruitment. Disease progression will be classified as a Y/N indicator in order to look at the proportion of those progressing in each cohort, using logistic regression to adjust for covariates of interest, such as age at diagnosis, tumour-node-metastasis stage, and Gleason score. Rate ratios for the cumulative incidence of disease progression for any disease, compared between the two cohorts, will be calculated using Poisson regression offset by person-years of follow-up, adjusting for covariates of interest.
To determine the incidence of aggressiveness of PrCa in the cohorts studied. | The full analysis being completed within one year of date of completion of 5 year follow-up of the last participant.
  Participants will be defined as experiencing disease progression if they have an upstaging or progression of their disease on MRI or biopsy. i.e., change in MRI or change in Gleason. Rate ratios for the cumulative incidence of aggressive disease (defined as progression on MRI or biopsy that results in the need for active treatment within one year of starting AS), compared between the two cohorts, will be calculated using Poisson regression offset by person-years of follow-up, adjusting for covariates of interest.

SECONDARY OUTCOMES:
To investigate the role of biomarker profiles in men undergoing active surveillance who are also at genetically higher risk for PrCa. | 5 years
  We will focus on DW-MRI at diagnosis, again using descriptive statistics and time-to-event analyses to break down the incidence of disease progression in each cohort and determine the association and interaction between higher genetic risk and DW-MRI.
To investigate the role of biomarker profiles in men undergoing active surveillance who are also at genetically higher risk for PrCa. | 5 years
  We will focus on metabolites using descriptive statistics and time-to-event analyses to break down the incidence of disease progression in each cohort and determine the association and interaction between higher genetic risk and metabolite levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ros A Eeles, FRCP, FRFR, Principal Investigator — Institute of Cancer Research and Royal Marsden Hospital
Locations (4):
- United Kingdom (4):
  - Institute of Cancer Research and Royal Marsden Hospital, Sutton, Surrey
  - North Bristol NHS Trust, Bristol
  - The Royal Marsden Hospital, London
  - The Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data can be applied for via the Data Access Committee

REFERENCES:
- [Background] Hamdy FC, Donovan JL, Lane JA, Mason M, Metcalfe C, Holding P, Davis M, Peters TJ, Turner EL, Martin RM, Oxley J, Robinson M, Staffurth J, Walsh E, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Neal DE; ProtecT Study Group. 10-Year Outcomes after Monitoring, Surgery, or Radiotherapy for Localized Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1415-1424. doi: 10.1056/NEJMoa1606220. Epub 2016 Sep 14. PMID 27626136
- [Background] Tseng KS, Landis P, Epstein JI, Trock BJ, Carter HB. Risk stratification of men choosing surveillance for low risk prostate cancer. J Urol. 2010 May;183(5):1779-85. doi: 10.1016/j.juro.2010.01.001. Epub 2010 Mar 20. PMID 20304433
- [Background] Bokhorst LP, Valdagni R, Rannikko A, Kakehi Y, Pickles T, Bangma CH, Roobol MJ; PRIAS study group. A Decade of Active Surveillance in the PRIAS Study: An Update and Evaluation of the Criteria Used to Recommend a Switch to Active Treatment. Eur Urol. 2016 Dec;70(6):954-960. doi: 10.1016/j.eururo.2016.06.007. Epub 2016 Jun 19. PMID 27329565
- [Background] Porten SP, Whitson JM, Cowan JE, Cooperberg MR, Shinohara K, Perez N, Greene KL, Meng MV, Carroll PR. Changes in prostate cancer grade on serial biopsy in men undergoing active surveillance. J Clin Oncol. 2011 Jul 10;29(20):2795-800. doi: 10.1200/JCO.2010.33.0134. Epub 2011 May 31. PMID 21632511
- [Background] Berglund RK, Masterson TA, Vora KC, Eggener SE, Eastham JA, Guillonneau BD. Pathological upgrading and up staging with immediate repeat biopsy in patients eligible for active surveillance. J Urol. 2008 Nov;180(5):1964-7; discussion 1967-8. doi: 10.1016/j.juro.2008.07.051. Epub 2008 Sep 17. PMID 18801515